CLINICAL TRIAL: NCT02714218
Title: Phase IIIb/IV, Randomized, Double Blinded, Study of Nivolumab 3 mg/kg in Combination With Ipilimumab 1 mg/kg vs Nivolumab 1 mg/kg in Combination With Ipilimumab 3 mg/kg in Subjects With Previously Untreated, Unresectable or Metastatic Melanoma
Brief Title: A Study of Two Different Dose Combinations of Nivolumab in Combination With Ipilimumab in Subjects With Previously Untreated, Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-511
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab 3 mg/kg IV; Biological: Ipilimumab 1 mg/kg IV
- Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab 1 mg/kg IV; Biological: Ipilimumab 3 mg/kg IV
- Nivolumab 6 mg/kg IV + Ipilimumab 1 mg/kg (Experimental): Specified dose on specified days
  Interventions: Biological: Ipilimumab 1 mg/kg IV; Biological: Nivolumab 6 mg/kg IV

INTERVENTIONS:
Biological: Nivolumab 3 mg/kg IV — Followed by Nivolumab monotherapy
  Arms: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV
Biological: Ipilimumab 1 mg/kg IV — Followed by Nivolumab monotherapy
  Arms: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV; Nivolumab 6 mg/kg IV + Ipilimumab 1 mg/kg
Biological: Nivolumab 1 mg/kg IV
  Arms: Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Biological: Ipilimumab 3 mg/kg IV
  Arms: Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Biological: Nivolumab 6 mg/kg IV — A dose of 240mg is identical to a dose of 3mg/kg, therefore 6mg/kg is approximately equal to ~ 480mg.
  Arms: Nivolumab 6 mg/kg IV + Ipilimumab 1 mg/kg

SUMMARY:
The purpose of this study is to evaluate two different dose combinations of nivolumab and ipilimumab in the treatment of melanoma.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subject must have been diagnosed with stage III or/and stage IV histologically confirmed melanoma [per American Joint Committee on Cancer (AJCC) staging system] that is unresectable or metastatic
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Subject has not been treated by systemic anticancer therapy for unresectable or metastatic melanoma

Exclusion Criteria:

* Subjects with active brain metastases or leptomeningeal metastases
* Subjects with ocular melanoma
* Subjects with active, known or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- United States (11):
  - University Of Colorado Cancer Center, Aurora, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Allina Health, Fridley, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University Of Virginia Health System, Charlottesville, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Local Institution, North Sydney, New South Wales
  - Local Institution - 0045, Waratah, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Melbourne, Victoria
- Canada (3):
  - Local Institution - 0007, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Quebec - Universite Laval, Québec, Quebec
- Denmark (3):
  - Local Institution - 0063, Aarhus N
  - Local Institution - 0065, Herlev
  - Local Institution - 0064, Odense
- France (8):
  - Hopital Saint Andre, Bordeaux
  - Chru De Lille, Lille
  - Hopital De La Timone, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Claudius Regaud, Toulouse
  - Local Institution - 0019, Villejuif
- Germany (4):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Ludwig-Maximilians-Universitaet, München
  - Universitaetsklinikum Tuebingen, Tübingen
- Local Institution, Ramat Gan, Israel
- Italy (6):
  - Local Institution - 0039, Bergamo
  - Local Institution - 0042, Milan
  - Local Institution - 0040, Napoli
  - Istituto Oncologico Veneto IOV, Padua
  - Local Institution - 0041, Siena
  - Ospedale San Vincenzo, Taormina
- Netherlands (3):
  - Local Institution - 0052, Amsterdam
  - Local Institution, Amsterdam
  - University Medical Center Groningen (Umcg), Groningen
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii I Radiote, Gdansk
  - Klinika Nowotworow Ukladowych i Uogolnionych, Krakow
  - Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- Local Institution, Moscow, Russia
- Spain (6):
  - Local Institution, Badalona-barcelona
  - Local Institution - 0024, Barcelona
  - Local Institution, Madrid
  - Local Institution - 0027, Madrid
  - Local Institution, San Sabastian Gipuzkoa
  - Local Institution, Valencia
- United Kingdom (4):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Oxford, Oxfordshire
  - Local Institution, Guildford
  - Local Institution, London

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Lebbe C, Meyer N, Mortier L, Marquez-Rodas I, Robert C, Rutkowski P, Menzies AM, Eigentler T, Ascierto PA, Smylie M, Schadendorf D, Ajaz M, Svane IM, Gonzalez R, Rollin L, Lord-Bessen J, Saci A, Grigoryeva E, Pigozzo J. Evaluation of Two Dosing Regimens for Nivolumab in Combination With Ipilimumab in Patients With Advanced Melanoma: Results From the Phase IIIb/IV CheckMate 511 Trial. J Clin Oncol. 2019 Apr 10;37(11):867-875. doi: 10.1200/JCO.18.01998. Epub 2019 Feb 27. PMID 30811280
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 387 participants were randomized, 385 were treated. Cohort C/N6I1 assessed for exploratory outcome measures not being reported in the Outcome Measures module. Safety data included with AE data.
Groups:
- Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV: nivolumab 3 mg/kg IV combined with ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then nivolumab (flat dose 480 mg) every 4 weeks.
- Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV: nivolumab 1 mg/kg IV combined with ipilimumab 3 mg/kg IV every 3 weeks for 4 doses then nivolumab (flat dose 480 mg) every 4 weeks
- Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg: nivolumab 6 mg/kg plus ipilimumab 1 mg/kg followed by nivolumab 480 mg Flat Dose 4 weeks later and repeated every 8 weeks
Period: Pre-Treatment Period
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg
Started | 180 | 180 | 27
Completed (Moved to treatment period) | 180 | 178 | 27
Not Completed | 0 | 2 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 0
Not completed — Other reasons | 0 | 1 | 0
Period: Treatment Period
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg
Started | 180 | 178 | 27
Completed | 6 | 2 | 2
Not Completed | 174 | 176 | 25
Not completed — Disease Progression | 55 | 52 | 14
Not completed — Study drug toxicity | 46 | 70 | 6
Not completed — Adverse event unrelated to study drug | 13 | 6 | 1
Not completed — Request to discontinue treatment | 1 | 4 | 1
Not completed — Participant withdrew consent | 2 | 2 | 0
Not completed — Maximum clinical benefit | 4 | 2 | 0
Not completed — Administrative reason by sponsor | 2 | 1 | 0
Not completed — Other reasons | 6 | 6 | 0
Not completed — Completed treatment as per protocol | 36 | 27 | 3
Not completed — Not reported | 9 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg | Total
Number analyzed (Participants) | 180 | 180 | 27 | 387
Age, Customized [Count of Participants; unit: Participants]
  <65 | 115 | 122 | 17 | 254
  >= 65 AND < 75 | 48 | 43 | 9 | 100
  >= 75 | 17 | 15 | 1 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 77 | 11 | 163
  Male | 105 | 103 | 16 | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 174 | 170 | 23 | 367
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Drug-Related Grade 3 - 5 Adverse Events (AEs)
Description: The percentage of participants who experienced at least 1 AE of Grade 3 or higher, judged to be related to study drug by the investigator, and with onset on or after the first dose of study treatment and within 30 days of the last dose of study treatment. AE grade was defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria.
Time Frame: From first dose of study treatment up to primary completion date 20-Apr-2017 (up to approximately 12 months)
Population: All treated participants in cohorts A and B
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 180 | 178
Percentage of participants | 32.8 [26.0 to 40.2] | 45.5 [38.0 to 53.1]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; p = 0.0144, Cochran-Mantel-Haenszel; Two-sided p-value CMH Test for comparison of odds ratio of NIVO 3 + IPI 1 over NIVO 1 + IPI 3; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.38 to 0.90]
Statistical Analysis 2: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; Estimated Difference of rates = -12.7, 95% CI 2-sided [-22.7 to -2.6] — Estimate of NIVO 3 + IPI 1- NIVO 1 + IPI 3 is based on Cochran-Mantel-Haenszel (CMH) method of weighting, adjusting for PD-L1 expression and M stage at screening as entered into the IVRS

2. Post Hoc Outcome: The Percentage of Participants With Drug-Related Grade 3 - 5 Adverse Events (AEs) - Extended Collection
Description: The percentage of participants who experienced at least 1 AE of Grade 3 or higher, judged to be related to study drug by the investigator, and with onset on or after the first dose of study treatment and within 30 days of the last dose of study treatment. AE grade was defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until study completion date: 28-May-2021)
Time Frame: From first dose of study treatment to 30 days after the last dose of study treatment (up to approximately 30 months)
Population: All treated participants in cohorts A and B
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 180 | 178
Percentage of participants | 33.9 [27.0 to 41.3] | 48.3 [40.8 to 55.9]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; p = 0.0059, Cochran-Mantel-Haenszel; Two-sided p-value CMH Test for comparison of odds ratio of NIVO 3 + IPI 1 over NIVO 1 + IPI 3; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.36 to 0.84]
Statistical Analysis 2: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; Estimated Difference of rates = -14.4, 95% CI 2-sided [-24.5 to -4.3] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). BOR is defined as the best response, as determined by the investigator, recorded between the date of randomization and the date of progression per RECIST 1.1 or the date of subsequent anticancer therapy, whichever occurred first. For subjects without documented progression or subsequent therapy, all available response designations will contribute to the BOR assessment. Tumor assessments are scheduled at Week 12 following randomization, every 8 weeks for the first 12 months and then every 12 weeks until disease progression. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization to date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (up to approximately 5 years)
Population: All treated participants in cohorts A and B
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 180 | 178
Percentage of participants | 47.8 [40.3 to 55.3] | 53.4 [45.8 to 60.9]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; p = 0.2923, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.53 to 1.21] — p-value from CMH Test for the comparison of the odds ratio of N3I1 over N1I3

4. Secondary Outcome: Overall Survival (OS)
Description: The time between the date of randomization and the date of death due to any cause. A participant who has not died will be censored at the last known alive date. OS will be followed continuously while participants are on the study drug and every 3 months via in-person or phone contact after participants discontinue the study drug. Based on Kaplan-Meier Estimates.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first (up tp approximately 5 years)
Population: All treated participants in cohorts A and B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 180 | 178
Months | NA [43.73 to NA] — Insufficient number of participants with events | NA [40.84 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.79 to 1.47] — Hazard Ratio is N3I1 over N1I3. (NIVO 3 + IPI 1 (N3I1) over NIVO 1 + IPI 3 (N1I3))

5. Secondary Outcome: Progression Free Survival (PFS)
Description: The time between the date of randomization and the first date of documented progression, determined by the investigator, or death due to any cause, whichever occurs first. Participants who die without a reported progression will be considered to have progressed on the date of their death. Those who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants without on study tumor assessments and who did not die will be censored on their date of randomization. Participants who started anti-cancer therapy without a prior reported progression will be censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy. Based on Kaplan-Meier Estimates. Progression is defined as at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to the first date of documented progression or death due to any cause, whichever occurs first (up to approximately 5 years)
Population: All treated participants in cohorts A and B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 180 | 178
Months | 10.18 [6.24 to 21.91] | 9.99 [6.28 to 28.88]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV vs Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV; Test type: Superiority; p = 0.4512, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.84 to 1.48]

6. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Physical Functioning Scale
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Physical Functioning Scale sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | -2.1 (16.2) | -4.9 (16.5)
  Week 16: number analyzed (Participants) | 63 | 47
  Week 16 | -1.9 (15.3) | -2.7 (15.8)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | -1.4 (10.7) | -2.7 (13.7)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -5.1 (15.6) | -5.7 (13.6)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | -2.5 (15.0) | -0.7 (14.8)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -3.3 (16.5) | -3.5 (15.4)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -4.0 (19.1) | -2.9 (14.8)
  Week 40: number analyzed (Participants) | 62 | 45
  Week 40 | -3.3 (17.3) | -3.4 (16.7)

7. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Role Functioning Scale
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Role Functioning Scale sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | -2.5 (28.3) | -8.8 (25.6)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | -6.6 (30.3) | 2.1 (25.6)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | -1.8 (19.9) | -5.2 (25.2)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -3.9 (19.9) | -9.8 (29.3)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | -0.9 (23.4) | -1.3 (26.0)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -3.6 (25.1) | -2.2 (29.3)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -3.9 (26.4) | -2.9 (30.5)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -4.0 (26.7) | -5.2 (34.2)

8. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Emotional Functioning Scale
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Emotional Functioning Scale sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 4.5 (17.9) | 4.4 (16.8)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 0.0 (21.7) | 6.6 (20.1)
  Week 20: number analyzed (Participants) | 72 | 58
  Week 20 | 3.9 (18.0) | 4.5 (18.0)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 3.4 (18.4) | 2.6 (23.3)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | 5.9 (19.5) | 5.6 (22.5)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 5.5 (17.3) | 5.1 (21.6)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 3.0 (17.0) | 4.7 (22.0)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 4.5 (21.4) | 5.4 (19.9)

9. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Cognitive Functioning Scale
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Cognitive Functioning Scale sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | -3.4 (15.0) | -1.9 (16.7)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | -2.6 (14.4) | -5.9 (22.4)
  Week 20: number analyzed (Participants) | 72 | 58
  Week 20 | -1.9 (16.9) | -6.0 (17.6)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -2.7 (15.0) | -3.4 (14.9)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | -3.7 (17.7) | -3.7 (16.8)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -1.5 (16.6) | -4.8 (16.9)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -3.1 (18.5) | -8.8 (20.6)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -2.6 (20.3) | -4.4 (15.2)

10. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Social Functioning Scale
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Social Functioning Scale sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 120 | 110
Scores on a scale
  Week 7 | -3.1 (22.8) | -6.1 (25.0)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | -6.3 (23.5) | -2.8 (26.7)
  Week 20: number analyzed (Participants) | 72 | 57
  Week 20 | -4.6 (21.0) | -3.2 (20.5)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -1.6 (17.2) | -3.7 (20.0)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | 1.4 (18.1) | -1.0 (22.2)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 0.3 (17.6) | -1.0 (19.6)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 0.5 (20.4) | 0.3 (22.7)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 1.1 (22.0) | -4.1 (23.3)

11. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Global Health Status
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The EORTC QLQ-C30 comprises 6 functional scales (role function, physical functioning, cognitive functioning, emotional functioning, social functioning and global quality of life) as well as nine symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). With the exception of 2 items included in the global health/quality of life scale, for which responses range from 1 (Very poor) to 7 (Excellent), item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores for all functional scales and Global Health Status indicate better HRQoL; an increase from baseline indicates improvement in HRQoL compared to baseline.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 120 | 111
Scores on a scale
  Week 7 | 0.5 (22.9) | -0.5 (19.0)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 0.0 (18.5) | 5.0 (24.5)
  Week 20: number analyzed (Participants) | 72 | 58
  Week 20 | -1.5 (19.9) | 0.0 (19.1)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -0.5 (16.1) | -1.6 (24.9)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | 0.7 (21.1) | 6.3 (23.4)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -0.5 (23.2) | 5.4 (23.9)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -2.9 (21.8) | 2.6 (25.6)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -0.8 (22.2) | 3.7 (21.1)

12. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Dyspnea
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Dyspnea sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 4.4 (21.5) | 6.3 (23.0)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 5.8 (22.0) | 2.1 (21.1)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | 2.7 (22.7) | 2.3 (22.4)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 2.3 (19.5) | 2.3 (22.4)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | 3.2 (25.7) | 0.0 (23.3)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 2.6 (23.1) | 2.6 (22.7)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 4.2 (21.8) | 0.0 (21.1)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 3.7 (22.5) | 2.2 (21.8)

13. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Insomnia
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Insomnia sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 120 | 112
Scores on a scale
  Week 7 | 0.6 (28.7) | -1.5 (30.5)
  Week 16: number analyzed (Participants) | 62 | 48
  Week 16 | -0.5 (28.0) | -2.8 (29.0)
  Week 20: number analyzed (Participants) | 72 | 58
  Week 20 | -0.9 (28.5) | -6.3 (28.9)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 2.3 (28.0) | -7.5 (26.5)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | 0.9 (25.6) | -7.3 (28.0)
  Week 32: number analyzed (Participants) | 65 | 51
  Week 32 | -3.1 (24.1) | -10.5 (29.4)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 0.5 (24.8) | -8.5 (30.4)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -1.1 (18.9) | -14.1 (31.4)

14. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Appetite Loss
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Appetite loss sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 3.0 (24.7) | 4.8 (28.6)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 2.1 (28.6) | -1.4 (31.5)
  Week 20: number analyzed (Participants) | 73 | 57
  Week 20 | 1.4 (21.8) | -3.5 (25.7)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -0.9 (22.9) | -2.9 (32.0)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | -0.9 (23.0) | -7.3 (26.3)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 1.0 (27.6) | -7.7 (23.4)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -2.6 (24.7) | -9.2 (26.7)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -2.6 (22.6) | -6.7 (31.5)

15. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Constipation
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Constipation sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 0.3 (26.4) | 2.4 (26.7)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 5.3 (22.6) | -2.8 (32.1)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | 3.7 (26.4) | 1.1 (25.7)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -0.5 (23.2) | -1.7 (26.8)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | 3.2 (27.5) | 1.4 (28.8)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 2.6 (23.1) | -5.1 (27.5)
  Week 36: number analyzed (Participants) | 63 | 51
  Week 36 | 3.7 (23.3) | -0.7 (29.4)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 1.1 (21.6) | 0.7 (29.7)

16. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Diarrhea
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Diarrhea sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points.
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 1.4 (18.5) | 1.2 (23.6)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 8.5 (22.4) | 2.8 (30.6)
  Week 20: number analyzed (Participants) | 72 | 58
  Week 20 | 2.3 (19.6) | -1.7 (22.0)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 1.8 (17.5) | 1.1 (25.7)
  Week 28: number analyzed (Participants) | 72 | 48
  Week 28 | 2.8 (19.2) | 0.0 (19.4)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 0.5 (19.1) | -2.6 (21.7)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 3.6 (16.9) | -2.0 (20.5)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -0.5 (18.4) | -3.7 (16.2)

17. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Financial Difficulties
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Financial difficulties sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 118 | 109
Scores on a scale
  Week 7 | 2.0 (24.4) | 2.4 (22.5)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 1.1 (19.8) | 4.9 (21.7)
  Week 20: number analyzed (Participants) | 72 | 57
  Week 20 | 2.8 (20.7) | 5.3 (19.7)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 1.8 (22.8) | 5.7 (17.8)
  Week 28: number analyzed (Participants) | 72 | 49
  Week 28 | 2.8 (23.6) | 6.8 (22.5)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 2.1 (22.7) | 5.8 (22.6)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 3.6 (22.3) | 8.5 (18.7)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 1.1 (23.9) | 8.1 (19.0)

18. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Fatigue
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Fatigue sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 5.1 (23.3) | 11.5 (23.2)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | 9.2 (25.8) | 5.1 (24.4)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | 4.4 (20.6) | 7.9 (20.5)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | 5.4 (20.5) | 6.9 (24.3)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | 4.8 (22.9) | 2.1 (19.5)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | 5.5 (23.7) | 3.2 (22.9)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 5.4 (27.1) | 1.7 (21.2)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 5.8 (24.3) | 0.7 (24.7)

19. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Nausea and Vomiting
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Nausea and Vomiting sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points for the various scales of the EORTC QLQ-C30
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 112
Scores on a scale
  Week 7 | 1.5 (16.4) | 4.9 (18.3)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | -0.3 (20.4) | 3.1 (11.7)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | -2.3 (10.1) | 1.1 (13.9)
  Week 24: number analyzed (Participants) | 73 | 58
  Week 24 | -0.5 (16.2) | 4.0 (18.0)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | 0.7 (13.5) | 0.7 (14.3)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -1.3 (14.2) | 0.3 (15.7)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | 0.0 (18.5) | 1.6 (16.1)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | -1.3 (12.1) | 0.7 (12.3)

20. Secondary Outcome: Mean Changes From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Pain
Description: Health Related Quality of Life (HRQoL) was assessed using the EORTC QLQ-C30 questionnaire. The Pain sub-scale item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores indicate a higher level of symptoms; lower scores indicating lesser burden and improved symptoms or quality of life. A clinically meaningful change in score may be regarded as 10 points
Time Frame: Weeks 7, 16, 20, 24, 28, 32, 36, 40
Population: All treated participants in cohorts A and B
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV
Number analyzed (Participants) | 121 | 111
Scores on a scale
  Week 7 | -1.7 (28.0) | 1.5 (25.6)
  Week 16: number analyzed (Participants) | 63 | 48
  Week 16 | -2.9 (22.9) | -2.8 (23.4)
  Week 20: number analyzed (Participants) | 73 | 58
  Week 20 | -5.7 (20.1) | 1.7 (28.0)
  Week 24: number analyzed (Participants) | 74 | 58
  Week 24 | -2.9 (20.9) | 0.9 (31.9)
  Week 28: number analyzed (Participants) | 72 | 50
  Week 28 | -3.0 (25.5) | -3.7 (30.9)
  Week 32: number analyzed (Participants) | 65 | 52
  Week 32 | -2.8 (27.1) | -4.5 (26.0)
  Week 36: number analyzed (Participants) | 64 | 51
  Week 36 | -2.6 (21.3) | -2.6 (29.9)
  Week 40: number analyzed (Participants) | 63 | 45
  Week 40 | 0.3 (25.3) | -3.3 (27.2)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events are collected from the first dose date until the last dose date + 30 days (Up to approximately 30 months) Participants were assessed for All Cause Mortality from their first dose until the study was completed (up to approximately 5 years)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg
All-Cause Mortality (participants affected / at risk) | 85/180 | 78/180 | 15/27
Serious Adverse Events (participants affected / at risk) | 109/180 | 127/178 | 14/27
Other Adverse Events (participants affected / at risk) | 169/180 | 172/178 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV (N=180) | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV (N=178) | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg (N=27)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 3 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 3 | 0
Hypophysitis (Endocrine disorders) | 2 | 6 | 1
Hypopituitarism (Endocrine disorders) | 0 | 2 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Orbital myositis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 6 | 10 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 12 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 2 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 3 | 1
Pyrexia (General disorders) | 5 | 11 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 5 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 4 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 8 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 3 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chorioretinitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0
Meningoencephalitis viral (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 4 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 3 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Spinal cord infection (Infections and infestations) | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Antibiotic level below therapeutic (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 3 | 0 | 0
Transaminases increased (Investigations) | 0 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 26 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Meningism (Nervous system disorders) | 0 | 0 | 1
Meningoradiculitis (Nervous system disorders) | 0 | 3 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Autoimmune nephritis (Renal and urinary disorders) | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg IV + Ipilimumab 1 mg/kg IV (N=180) | Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV (N=178) | Cohort C, Nivolumab 6 mg/kg + Ipilimumab 1 mg/kg (N=27)
Anaemia (Blood and lymphatic system disorders) | 20 | 17 | 4
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 3
Adrenal insufficiency (Endocrine disorders) | 4 | 12 | 1
Hyperthyroidism (Endocrine disorders) | 20 | 31 | 3
Hypophysitis (Endocrine disorders) | 10 | 12 | 3
Hypothyroidism (Endocrine disorders) | 27 | 41 | 2
Vision blurred (Eye disorders) | 6 | 9 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 36 | 25 | 6
Abdominal pain upper (Gastrointestinal disorders) | 12 | 16 | 2
Constipation (Gastrointestinal disorders) | 25 | 31 | 3
Diarrhoea (Gastrointestinal disorders) | 66 | 73 | 11
Dry mouth (Gastrointestinal disorders) | 16 | 28 | 3
Nausea (Gastrointestinal disorders) | 41 | 49 | 9
Vomiting (Gastrointestinal disorders) | 28 | 34 | 4
Asthenia (General disorders) | 49 | 54 | 8
Chills (General disorders) | 12 | 10 | 3
Fatigue (General disorders) | 66 | 51 | 8
Influenza like illness (General disorders) | 14 | 15 | 1
Mucosal inflammation (General disorders) | 2 | 6 | 2
Oedema peripheral (General disorders) | 18 | 12 | 2
Pyrexia (General disorders) | 39 | 47 | 6
Cholestasis (Hepatobiliary disorders) | 1 | 4 | 2
Hepatic cytolysis (Hepatobiliary disorders) | 6 | 6 | 3
Nasopharyngitis (Infections and infestations) | 16 | 16 | 5
Upper respiratory tract infection (Infections and infestations) | 14 | 8 | 1
Urinary tract infection (Infections and infestations) | 5 | 13 | 1
Alanine aminotransferase increased (Investigations) | 22 | 36 | 6
Amylase increased (Investigations) | 16 | 14 | 4
Aspartate aminotransferase increased (Investigations) | 18 | 30 | 5
Blood alkaline phosphatase increased (Investigations) | 10 | 3 | 2
Blood cholesterol increased (Investigations) | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 7 | 3 | 3
Blood creatinine increased (Investigations) | 6 | 12 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 1 | 2
Blood magnesium decreased (Investigations) | 0 | 0 | 2
Blood thyroid stimulating hormone decreased (Investigations) | 3 | 5 | 2
Blood thyroid stimulating hormone increased (Investigations) | 5 | 2 | 4
Cortisol decreased (Investigations) | 3 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 13 | 8 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 2
Lipase increased (Investigations) | 17 | 20 | 3
Neutrophil count decreased (Investigations) | 1 | 2 | 2
Protein total decreased (Investigations) | 0 | 1 | 2
Weight decreased (Investigations) | 25 | 29 | 1
Decreased appetite (Metabolism and nutrition disorders) | 37 | 31 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 17 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 9 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 36 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 23 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 10 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 15 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 16 | 5
Dizziness (Nervous system disorders) | 9 | 9 | 6
Headache (Nervous system disorders) | 38 | 51 | 4
Paraesthesia (Nervous system disorders) | 9 | 16 | 1
Anxiety (Psychiatric disorders) | 7 | 7 | 2
Insomnia (Psychiatric disorders) | 24 | 18 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 35 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 26 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 11 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 7 | 5 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 55 | 60 | 13
Rash (Skin and subcutaneous tissue disorders) | 42 | 54 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 7 | 8 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 17 | 5
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 21 | 16 | 3
Hypertension (Vascular disorders) | 9 | 6 | 3
Lymphoedema (Vascular disorders) | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02714218/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02714218/SAP_001.pdf